CLINICAL TRIAL: NCT02127931
Title: Predictive Executive Functioning Models Using Interactive Tangible-Graphical Interface Devices in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CogCubed, Corp (Industry)
Responsible Party: Principal Investigator, Monika Roots, MD, CogCubed, Corp
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NCT01711372B
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Video Game Diagnostic Tool Groundskeeper, a Video Game Diagnostic Tool for ADHD is administer to probands with ADHD and age, gender matched controls without ADHD.
Who Masked: Participant, Investigator
Masking Description: The participant does not know if they have ADHD symptoms or not and the investigator who is administering the game does not know what group the patient is in.
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADHD group played Game (Experimental): Groundskeeper, a Video Game Diagnostic Tool for ADHD is administer to probands with ADHD and age, gender matched controls without ADHD. The game was played on Sifteo cubes.
  Interventions: Device: Groundskeeper for ADHD group
- Control group played game (Active Comparator): Groundskeeper, a Video Game Diagnostic Tool for ADHD is administer to probands with ADHD and age, gender matched controls without ADHD. The game was played on Sifteo cubes.
  Interventions: Device: Groundskeeper for control group

INTERVENTIONS:
Device: Groundskeeper for ADHD group — Groundskeeper, a Video Game Diagnostic Tool for ADHD is administered to probands with ADHD and age, gender matched controls without ADHD.
  Arms: ADHD group played Game
Device: Groundskeeper for control group — Groundskeeper, a Video Game Diagnostic Tool for ADHD is administered to probands with ADHD and age, gender matched controls without ADHD.
  Arms: Control group played game

SUMMARY:
Current diagnostic aids used in treating ADHD are currently expensive, time intensive, and provide little information about accessory movements in response to a stimulus.

Tests such as the Conners' Rating Scale require subjective responses from parents and teachers, making coordination difficult. The computerized Conners' Continuous Performance Test (CPT) provides objective data in regards to inattention and impulsive patterns of response. However, it does not provide data regarding accessory movements such as restlessness, hyperactivity, and other inappropriate movements. If the subject taking the exam has a reading disorder, it will impair his or her ability to respond accurately and it will increase response time. The T.O.V.A. is another computer based test used as a diagnostic aid for ADHD, which uses a microswitch to record responses. It does utilize auditory and visual stimuli, which removes the reading level limitation. However, it is unable to measure to measure accessory movements that may be contributing to reaction time and errors of omission and commission.

Because of these limitations, a new company called CogCubed has created a new game based on the Sifteo Cube (http://www.sifteo.com) platform. These new hands-on digitized cubes are unique, motion-sensitive wireless blocks that contain multiple sensors that can interact with one another. CogCubed is providing the data for this study. The game will be played in a 30 minute sessions by subjects aged 18 and over. Subjects recruited to play the game will be those with ADHD and those without, matched by gender. Those with comorbidities of developmental delay, mental retardation, psychosis, schizophrenia, bipolar disorder and substance use disorders will be excluded, as well as any physiological disability that affects upper limb movement and/or coordination. Informed consent will be obtained from participant prior to administering the game.

The hypothesis is that by analyzing data generated from this new gaming platform named Sifteo for which a game was created, which uses auditory and visual stimuli and distracters, the investigators expect that they will be able to provide a more accurate profile of impulsivity and inattention. The investigators expect that inattention will have more errors of omission and less tilt movements than control and impulsivity will be represented as more commission and greater tilting movements than control.

DETAILED DESCRIPTION:
This trial builds on the previous results of our phase 1 trials in children ages 6-17 used to create the predictive algorithms to analyze the data and predict the likelihood of ADHD diagnosis based on patterns of game play behavior. Participants in this study will complete the Schedule for Affective Disorders and Schizophrenia (SADS), the DSM IV Adult ADHD Checklist, Hamilton Rating Scal for Depression (HRSD), the Hamilton Rating Scale for Anxiety (HAM-A), and complete the Conner's Continuous Performance test (CPT 3).

ELIGIBILITY:
Inclusion Criteria:

* Age 18+, males and females
* Individuals with ADHD
* Individuals without ADHD
* Depressive Disorders
* Anxiety Disorders
* High functioning Autism Spectrum Disorders
* Mood Disorders

Exclusion Criteria:

* Under the age of 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Roots, MD, Principal Investigator — CogCubed, Corp
Locations (1):
- Macalester College, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a highly selective college
Pre-assignment Details: Company no longer exists, and no longer has access to data collected. Only information from draft publication available.
Groups:
- All Participants: College students recruited for study Groundskeeper: Groundskeeper, a Video Game Diagnostic Tool for ADHD is administered to probands with ADHD and age, gender matched controls without ADHD.
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 17
Not Completed | 1
Not completed — Glitch in Game | 1

BASELINE CHARACTERISTICS:
Population: Company no longer exists, and no longer has access to data collected. Only information from draft publication available.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 18
Sex/Gender, Customized [Count of Participants; unit: Participants] — Information of Sex/Gender is unknown as information is not available for analysis
  Participants
    NA | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — N/A, Information is not available for analysis and is not information is unknown.
  Participants
    N/A | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Tested High (6 or More Symptoms) for ADHD by Type Determined by Adult ADHD DSM IV-TR Checklist
Description: Adult ADHD DSM IV-TR Checklist for determining ADHD subtypes: inattentive ADHD (ADHD-I), Hyperactive/impulsive ADHD (ADHD-H/I) and Combined ADHD (ADHD-C). Company no longer exitsts, and no longer has access to data collected. Only information from draft publication available
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 17
Participants
  ADHD- H/I | 2
  ADHD-I | 5
  ADHD-C | 2

2. Primary Outcome: Correlation of CPT Commission Errors With ADHD-I and ADHD-C
Description: Continuous performance task (CPT), participants are asked to press the space bar when they are presented with any letter except the letter "X". The participant must refrain from clicking if they see the letter "X" presented.
Time Frame: 14 minutes
Measure: Number; unit: Correlation
Groups:
- All Participants: College students and participants requested to complete CPT
Arm/Group | All Participants
Number analyzed (Participants) | 17
Correlation
  ADHD-I | 0.648
  ADHD-C | 0.587
Statistical Analysis 1: Comparison: All Participants; ADHD-I; Test type: Other; p = 0.005, Correlation
Statistical Analysis 2: Comparison: All Participants; ADHD-C; Test type: Other; p = 0.023, Correlation

3. Primary Outcome: Correlation of Groundskeeper Incorrect With CPT Commission Errors
Description: Groundskeeper is a game, there are four cubes and a base device, three of the cubes display a background of a grassy field, with occasional stimuli that pop up. The fourth cube displays a mallet. When a gopher is displayed on one of the cubes, the user must hit the gopher with the mallet. Groundskeeper incorrect counts of the number of incorrect responses when a target stimulus is presented. Continuous performance task (CPT), participants are asked to press the spacebar each time a letter appears in the middle of the screen, except when the letter is "X." If the letter is an "X", the participant should do nothing. Commission errors were when participant pressed the spacebar when an "X" appeared. Company no longer exists, and no longer has access to data collected. Only information from draft publication available.
Time Frame: 45 minutes
Measure: Number; unit: Correlation
Arm/Group | All Participants
Number analyzed (Participants) | 17
Correlation | 0.587
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.013, Correlation

ADVERSE EVENTS:
Description: Company no longer exists, and no longer has access to data collected. Only information from draft publication available. No information available on monitoring/frequency of Adverse Events
Groups:
- College Students and Participants Requested to Complete CPT: Groundskeeper, a Video Game Diagnostic Tool for ADHD is administer to probands with ADHD and age, gender matched controls without ADHD.
  Groundskeeper for ADHD group: Groundskeeper, a Video Game Diagnostic Tool for ADHD is administered to probands with ADHD and age, gender matched controls without ADHD.
Arm/Group | College Students and Participants Requested to Complete CPT
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes